CLINICAL TRIAL: NCT03147742
Title: An Open-Label, Expanded Access Program of Ruxolitinib for the Treatment of Graft-Versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: An Expanded Access Program of Ruxolitinib for the Treatment of Graft-Versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplant
Status: Approved for marketing | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB 18424-MA-GD-301
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: ruxolitinib; acute or chronic steroid-refractory GVHD; hematopoietic stem cell transplantation (allo-HSCT)
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib starting dose level 10 mg orally, twice daily (BID).
  Other Names: INCB018424

SUMMARY:
To provide ruxolitinib through an expanded access program for the treatment of graft-versus-host disease (GVHD) in United States to patients who are ineligible or unable to participate in any actively enrolling Incyte-sponsored clinical studies for ruxolitinib in the treatment of GVHD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 12 years of age or older.
* Have undergone an allo-HSCT from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative conditioning regimens are eligible.
* Clinically suspected all grades chronic GVHD according to NIH Consensus Criteria that is refractory or intolerant to corticosteroids, occurring after allo-HSCT with any conditioning regimen and any anti-GVHD prophylactic regimen. Clinical suspicion of steroid-refractory chronic GVHD by the treating physician is also sufficient.
* Evidence of myeloid engraftment (eg, absolute neutrophil count ≥ 1.0 × 10^9/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
* Evidence of platelet engraftment (ie, platelets ≥ 20 × 10^9/L).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3.
* Be willing to avoid pregnancy or fathering children based on 1 of the following criteria:

  * Women of non-childbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea).
  * Woman of childbearing potential who has a negative serum pregnancy test at screening and who agrees to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the patient and their understanding confirmed.
  * Man who agrees to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the patient and their understanding confirmed.
* Able to provide written informed consent and/or assent from the patient, parent, or guardian.

Key Exclusion Criteria:

* Eligible for an existing and actively enrolling Incyte sponsored clinical trial for ruxolitinib for the treatment of GVHD.
* Clinically suspected all grades of acute GVHD as per Minnesota-Center for International Blood and Marrow Transplant Research (MN-CIBMTR) criteria or clinical suspicion of acute GVHD by the treating physician.
* Patients or legal guardians unable to review and sign informed consent form.
* Females who are pregnant or breastfeeding, and males and females who cannot comply with requirements to avoid fathering a child or becoming pregnant.
* Patients with inadequate liver function (alanine aminotransferase above 4 × upper limit of normal (ULN) or direct bilirubin 4 × ULN and the laboratory abnormalities are considered to be due to underlying liver dysfunction) unless attributed to GVHD.
* Patients with end stage renal function (creatinine clearance (CrCl) < 15 mL/min or glomerular filtration rate < 15 mL/min), regardless of whether hemodialysis is required.
* Any underlying or current medical or psychiatric condition that, in the opinion of the treating physician, would place the patient at an unacceptable risk if he or she were to participate in the program.
* Previous allergic reactions to Janus kinase (JAK) inhibitors or excipients.
* Patients who are currently taking any anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, or tumor embolization).
* Concomitant use of any JAK inhibitor.
* Initiating therapy with any investigational medication.
* Presence of an active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Known HIV infection.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Previous test results obtained as part of standard of care before allo-HSCT that confirm a patient is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Galvin, MD, Study Director — Incyte Corporation
Locations (33):
- United States (33):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cancer Transplant Institute at HonorHealth, Scottsdale, Arizona
  - City of Hope Medical Center, Duarte, California
  - Scripps Clinic, La Jolla, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Blood & Marrow Transplant Center, Orlando, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Allegheny Health Network Cancer Institute, Pittsburgh, Pennsylvania
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Texas Oncology, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin